CLINICAL TRIAL: NCT02679287
Title: Project Nightlight: Efficacy and System Acceptance of Dinner/Night vs. 24hr Closed Loop Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Roche Diagnostic Ltd. (Industry); TypeZero Technologies, LLC (Industry); Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Sue Brown, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18617; R01DK085623 (NIH)
Record Dates: First submitted 2016-01-08; First posted 2016-02-10 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Closed-Loop Control (CLC); Sensor-Augmented Therapy (SAP); USS Virginia; Continuous Glucose Monitor (CGM); Insulin Pump; Artificial Pancreas (AP)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group A (Experimental): Order of intervention will be 1) SAP; 2) USS + SAP(d); 3) USS +CLC (d); 4) USS + SAP(d)
  1. SAP=sensor-augmented pump only
  2. USS+SAP (d)= Evening and Overnight Closed-Loop Control=SAP during day and CLC starting at dinner and continuing overnight
  3. USS+CLC (d)= 24/7 Closed-Loop Control=24-hour Day and Night Closed Loop Control
  Interventions: Device: CLC
- Group B (Experimental): Order of intervention will be 1)USS + SAP(d) ; 2)USS +CLC (d); 3) USS + SAP(d); 4) SAP
  1. SAP=sensor-augmented pump only
  2. USS+SAP (d)= Evening and Overnight Closed-Loop Control=SAP during day and CLC starting at dinner and continuing overnight
  3. USS+CLC (d)= 24/7 Closed-Loop Control=24-hour Day and Night Closed Loop Control
  Interventions: Device: CLC

INTERVENTIONS:
Device: CLC — The CLC will be deployed with different functionalities at different stages of the trial, resulting in variation in what the subject will be responsible for and what the system will drive.
  Other Names: Closed Loop Control

SUMMARY:
The purpose of this study is to use an investigational type of technology called Closed-Loop Control (CLC) Medical Platform System to help control blood sugar in people with type 1 diabetes mellitus in a home setting.

DETAILED DESCRIPTION:
The CLC is an "artificial pancreas" (AP) application that uses advanced closed loop control algorithms to automatically manage blood glucose levels for people with Type 1 Diabetes. The system modulates insulin to keep blood glucose in a targeted range. The CLC will be deployed with different functionalities at different stages of the trial, resulting in variation in what the subject will be responsible for and what the system will drive.These functionalities occur in a randomized cross-over design, each occurring for 8 weeks. These modalities are:

1. SAP=sensor-augmented pump only
2. USS+SAP (d)= Evening and Overnight Closed-Loop Control=SAP during day and CLC starting at dinner and continuing overnight
3. USS+CLC (d)= 24/7 Closed-Loop Control=24-hour Day and Night Closed Loop Control

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes for at least one year
* using insulin for at least 1 year
* an insulin pump for at least 6 months
* willingness to switch to lispro (Humalog) or aspart (Novolog) if using glulisine (Apidra).

Exclusion Criteria:

* a medical condition or being been treated with medications that might interfere with the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-02; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue A. Brown, MD, Principal Investigator — UVA Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Generally will be available after publications completed.

REFERENCES:
- [Derived] Kovatchev BP, Kollar L, Anderson SM, Barnett C, Breton MD, Carr K, Gildersleeve R, Oliveri MC, Wakeman CA, Brown SA. Evening and overnight closed-loop control versus 24/7 continuous closed-loop control for type 1 diabetes: a randomised crossover trial. Lancet Digit Health. 2020 Feb;2(2):e64-e73. doi: 10.1016/S2589-7500(19)30218-3. Epub 2020 Jan 3. PMID 32864597

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 103 participants signed informed consent and were assessed for eligibility.10 were excluded prior to randomization (7 did not meet inclusion criteria, 2 declined to participate, 1 lost to followup). 93 participants were randomized and assigned to groups.
Groups:
- Group A: Order of intervention will be 1) SAP; 2) USS + SAP(d); 3) USS +CLC (d); 4) USS + SAP(d)
  CLC: The CLC will be deployed with different functionalities at different stages of the trial, resulting in variation in what the subject will be responsible for and what the system will drive.
  1. SAP=sensor-augmented pump only
  2. USS+SAP (d)= Evening and Overnight Closed-Loop Control=SAP during day and CLC starting at dinner and continuing overnight
  3. USS+CLC (d)= 24/7 Closed-Loop Control=24-hour Day and Night Closed Loop Control
- Group B: Order of intervention will be 1)USS + SAP(d) ; 2)USS +CLC (d); 3) USS + SAP(d); 4) SAP
  CLC: The CLC will be deployed with different functionalities at different stages of the trial, resulting in variation in what the subject will be responsible for and what the system will drive.
  1. SAP=sensor-augmented pump only
  2. USS+SAP (d)= Evening and Overnight Closed-Loop Control=SAP during day and CLC starting at dinner and continuing overnight
  3. USS+CLC (d)= 24/7 Closed-Loop Control=24-hour Day and Night Closed Loop Control
Period: Period 1: Randomization-Study Session 1
Arm/Group | Group A | Group B
Started (Randomization) | 47 | 46
Completed (Completion of Study Session 1 Group A=SAP Group B=Evening/Overnight CLC) | 43 | 40
Not Completed | 4 | 6
Not completed — Regimen not compatible with study | 2 | 1
Not completed — Work or scheduling conflict | 2 | 3
Not completed — Disliked mobile system | 0 | 1
Not completed — Adverse Event prior to intervention | 0 | 1
Period: Period 2
Arm/Group | Group A | Group B
Started | 43 | 40
Completed (Completed Study Session 2: Group A: Evening/Overnight CLC Group B: 24/7 CLC) | 40 | 40
Not Completed | 3 | 0
Not completed — Work/Scheduling Conflict | 1 | 0
Not completed — Disliked Mobile System | 2 | 0
Period: Period 3
Arm/Group | Group A | Group B
Started | 40 | 40
Completed (Completed Study Session 3: Group A: 24/7 CLC Group B: Evening/Overnight CLC) | 40 | 39
Not Completed | 0 | 1
Not completed — Work/Scheduling Conflict | 0 | 1
Period: Phase 4
Arm/Group | Group A | Group B
Started (Completed Study Session 4: Group A: Evening/Overnight CLC Group B: SAP) | 40 | 39
Completed | 40 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analyzed group includes participants who completed two study sessions or more.
Groups:
- Group A: Order of intervention will be 1) SAP; 2) USS + SAP(d); 3) USS +CLC (d); 4) USS + SAP(d)
  CLC: The CLC will be deployed with different functionalities at different stages of the trial, resulting in variation in what the subject will be responsible for and what the system will drive.
- Group B: Order of intervention will be 1)USS + SAP(d) ; 2)USS +CLC (d); 3) USS + SAP(d); 4) SAP
  CLC: The CLC will be deployed with different functionalities at different stages of the trial, resulting in variation in what the subject will be responsible for and what the system will drive.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (13.5) | 41.9 (10.1) | 42.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 13 | 14 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/More than One Race | 38 | 40 | 78
  Asian | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Hemoglobin A1c [Mean (Standard Deviation); unit: percent] | 7.6 (1.08) | 7.24 (0.97) | 7.42 (1.03)

OUTCOME MEASURES:

1. Primary Outcome: Time <70 mg/dl by CGM
Description: Overnight CLC achieved by USS+SAP(d) (also known at Evening-Night CLC) will be superior to SAP alone in terms of reduced incidence and risk for hypoglycemia overnight without deterioration in hemoglobin A1c. Outcomes will be stratified by Hemoglobin A1c < 7.5% vs ≥7.5% and time of day.
Time Frame: 8 weeks
Population: This primary analysis was confined to the phase of the study comparing SAP to Evening-Night CLC only when combining group A and B. Data on 24/7 CLC phase is included in secondary outcomes.
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Group A and Group B Combined: Order of interventions for Group A 1) SAP; 2) USS + SAP(d); 3) USS +CLC (d); 4) USS + SAP(d)
  Order of intervention for Group B 1)USS + SAP(d) ; 2)USS +CLC (d); 3) USS + SAP(d); 4) SAP
  SAP=Sensor-augmented pump (study CGM+personal pump) USS+SAP(d)=Evening-Overnight CLC USS+CLC= 24/7 CLC
  CLC: The CLC will be deployed with different functionalities at different stages of the trial, resulting in variation in what the subject will be responsible for and what the system will drive.
Arm/Group | Group A and Group B Combined
Number analyzed (Participants) | 78
percentage of time
  CGM Time<70 mg/dL in SAP | 4.0 (3.3)
  CGM Time<70 mg/dL in Evening-Overnight CLC | 2.2 (1.8)
Statistical Analysis 1: Comparison: Group A and Group B Combined; The null hypothesis is that there is no difference in percentage of time <70 mg/dL in SAP vs. evening-overnight CLC session. Change in HbA1c during study sessions was used as a covariate of the model; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [1.2 to 2.4]

2. Primary Outcome: Hemoglobin A1c
Description: Overnight CLC achieved by USS+SAP(d) (also known as Evening-Night CLC) will be superior to SAP alone in terms of reduced incidence and risk for hypoglycemia overnight without deterioration in hemoglobin A1c. Outcomes will be stratified by Hemoglobin A1c < 7.5% vs ≥7.5% and time of day.
Time Frame: 8 weeks
Population: This primary analysis was confined to the phase of the study comparing SAP to Evening-Night CLC only when combining group A and B and included the baseline HbA1c and final HbA1c. Data on HbA1c by study phase is included in secondary outcomes.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Group A and Group B Combined
Number analyzed (Participants) | 78
percentage of glycated hemoglobin
  HbA1c at baseline | 7.42 (1.03)
  HbA1c at end of study | 7.11 (0.86)

3. Secondary Outcome: Time Between 70-180 mg/dL by CGM
Description: Time in target range 70-180 mg/dL measured by CGM
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Sensor-augmented Pump Therapy (SAP): Use of study CGM and personal pump for 8 weeks.
- Evening and Overnight Closed-Loop Control: Use of CLC evening to overnight hours for two sessions of 8 weeks
- 24/7 Closed-Loop Control: Use of CLC 24/7 for 8 weeks
Arm/Group | Sensor-augmented Pump Therapy (SAP) | Evening and Overnight Closed-Loop Control | 24/7 Closed-Loop Control
Number analyzed (Participants) | 77 | 77 | 77
percentage of time | 58.6 (14.6) | 67.6 (12.9) | 69.5 (10.9)

4. Secondary Outcome: Time >180 mg/dL by CGM
Description: Time in hyperglycemia range >180 mg/dL measured by CGM
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Sensor-augmented Pump Therapy (SAP) | Evening and Overnight Closed-Loop Control | 24/7 Closed-Loop Control
Number analyzed (Participants) | 77 | 77 | 77
percentage of time | 37.4 (16.5) | 30.1 (13.7) | 28.7 (11.4)

5. Secondary Outcome: Mean Glucose by CGM
Description: Mean glucose measured by CGM overall in mmol/L
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sensor-augmented Pump Therapy (SAP) | Evening and Overnight Closed-Loop Control | 24/7 Closed-Loop Control
Number analyzed (Participants) | 77 | 77 | 77
mmol/L | 9.3 (1.58) | 8.82 (1.22) | 8.74 (0.99)

6. Secondary Outcome: Low Blood Glucose Index (LBGI)
Description: Index measure of low blood glucose risk. This is an index that indicates risk of hypoglycemia with low values indicating lower risk of hypoglycemia (particularly values 1 or lower).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Sensor-augmented Pump Therapy (SAP) | Evening and Overnight Closed-Loop Control | 24/7 Closed-Loop Control
Number analyzed (Participants) | 77 | 77 | 77
index | 1.04 (0.79) | 0.66 (0.42) | 0.57 (0.34)

7. Secondary Outcome: High Blood Glucose Index (HBGI)
Description: Index measure of high blood glucose risk.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Sensor-augmented Pump Therapy (SAP) | Evening and Overnight Closed-Loop Control | 24/7 Closed-Loop Control
Number analyzed (Participants) | 77 | 77 | 77
index | 8.82 (4.61) | 6.97 (3.52) | 6.53 (2.86)

8. Secondary Outcome: CGM <70mg/dL
Description: Percentage time <70mg/dL measured by CGM in three study phases combining Group A and B.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Sensor-augmented Pump Therapy (SAP) | Evening and Overnight Closed-Loop Control | 24/7 Closed-Loop Control
Number analyzed (Participants) | 77 | 77 | 77
Percentage of time | 4.0 (3.3) | 2.3 (1.7) | 1.8 (1.4)

9. Secondary Outcome: Hemoglobin A1c by Study Session
Description: Hemoglobin A1c after each 8 weeks study session by Group A and Group B.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Group A | Group B
Number analyzed (Participants) | 40 | 40
percentage of glycated hemoglobin
  Session 1 (Group A SAP; Group B evening-night CLC) | 7.3 (0.83) | 7.01 (0.76)
  Session 2 (Gp A Evening-NIght CLC;Gp B 24/7 CLC) | 7.12 (0.79) | 6.95 (0.68)
  Session 3 (Gp A 24/7 CLC; Gp B evening-night CLC | 7.13 (0.8) | 7.06 (0.95)
  Session 4 (Gp A Evening-Night CLC; Gp B SAP) | 7.1 (0.73) | 7.12 (0.97)

ADVERSE EVENTS:
Time Frame: Approximately 10-11 months.
Groups:
- Sensor-Augmented Pump Therapy (SAP); 24/7 Closed-Loop Control: 8 week study phase for both Group A and Group B that underwent the same procedures in different orders.
- Evening and Overnight Closed-Loop Control: 8 week study phases (2) for both Group A and Group B that underwent the same procedures in different orders.
- Other: This includes any study periods outside of other study phases listed such as screening and washout periods for both Group A and Group B that underwent the same procedures in different orders.
Arm/Group | Sensor-Augmented Pump Therapy (SAP) | Evening and Overnight Closed-Loop Control | 24/7 Closed-Loop Control | Other
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/93 | 0/93 | 0/93
Serious Adverse Events (participants affected / at risk) | 1/93 | 1/93 | 0/93 | 1/93
Other Adverse Events (participants affected / at risk) | 5/93 | 14/93 | 7/93 | 9/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensor-Augmented Pump Therapy (SAP) (N=93) | Evening and Overnight Closed-Loop Control (N=93) | 24/7 Closed-Loop Control (N=93) | Other (N=93)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip Replacement Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Cell Carcinoma with Surgical Resection (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensor-Augmented Pump Therapy (SAP) (N=93) | Evening and Overnight Closed-Loop Control (N=93) | 24/7 Closed-Loop Control (N=93) | Other (N=93)
Severe Hypoglycemia (Endocrine disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) — Hypoglycemia requiring the assistance of a third party.
Hyperglycemia with ketosis not meeting diabetes ketoacidosis criteria (Endocrine disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) — Significantly elevated ketones requiring intervention without meeting DCCT criteria for diabetic ketoacidosis
Trauma (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Infections requiring medications or interventions (Infections and infestations) | 4 (4) | 5 (5) | 2 (2) | 1 (1)
Conditions requiring steroid use (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) — e.g. cervical radiculopathy, knee injury, tenosynovitis, dermatitis
Outpatient surgery or procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
New onset Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burn (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
New onset edema requiring medications (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT02679287/Prot_SAP_ICF_000.pdf